CLINICAL TRIAL: NCT00853060
Title: Energy Expenditure During Weaning From Mechanical Ventilation: Is There Any Difference Between Pressure Support and T-Tube?
Brief Title: Energy Expenditure in Weaning From Mechanical Ventilation
Status: Completed | Type: Observational
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Silvia Regina Rios Vieira, Hospital de Clínicas de Porto Alegre
Other Study IDs: 04-415
Record Dates: First submitted 2009-02-25; First posted 2009-02-27 (Estimated); Last update posted 2009-02-27 (Estimated); Status verified 2009-02

CONDITIONS: Respiration, Artificial; Energy Metabolism
Keywords: energy expenditure; mechanical ventilation; weaning; pressure support ventilation; T-tube
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
During weaning from mechanical ventilation process, the energy expenditure in T tube is greater than pressure support ventilation.

DETAILED DESCRIPTION:
The energy expenditure (EE) was measured during the two periods of 30-minutes, with the 10 first minutes being discarded for analysis purposes. The other variables were recorded and monitored during the 10th and the 30th minute, in both pressure support (PS) and t-Tube (TT) modes. Patients were randomized in terms of sequence selection: PS - TT or TT - PS. In the baseline period, patients were receiving mechanical ventilation (Servo 900C and Servo 300; Siemens-Elema, Solna, Sweden), with PS ranging from 10 to 15cmH2O. During the PS mode, patients received assisted pressure ventilation of 10 cmH2O, 5 cmH2O of final positive expiratory pressure, the sensitivity of -1cmH2O and FiO2 of 0.4. During TT mode, oxygen flow was delivered in order to keep the same FiO2 that was provided in PS (0.4) as controlled by monitor screen (Datex Ohmeda S/5 - Compact Airway Module, M-COVX model, Finland). In this mode, an extensor was employed, one end of which was connected to the oxygen-enriched and the other end was secured to a 3-output ("T") connector, which was attached to the patient's ventilatory prosthesis. During the rest period (30 minutes), patients returned to the mechanical ventilation parameters utilized in the baseline period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute respiratory failure receiving MV for over 24 hours, in the ICU of the Hospital de Clínicas de Porto Alegre

Exclusion Criteria:

* Patients with chest drainage, hemodynamic instability (characterized by the use of vasoactive drugs), renal failure, mental status change, agitation, sudoresis, tachycardia, axillary temperature above 38°C and inspiratory oxygen fraction (FiO2) over 0.6.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with respiratory failure receiving MV fore more than 24 hours, who had been admitted to the Intensive Care Unit (ICU) of the Hospital de Clínicas de Porto Alegre and who met the criteria for weaning from MV according to the parameters previously defined were selected to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Vieira, PhD, Principal Investigator — Federal University of Rio Grande do Sul
Locations (1):
- Federal University of Rio Grande do Sul/Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil